CLINICAL TRIAL: NCT05621369
Title: Psorcast Study: A Smartphone-based Study of Psoriasis and Psoriatic Arthritis
Brief Title: Psorcast Mobile Study
Status: Recruiting | Type: Observational
Sponsor: Sage Bionetworks (Other)
Collaborators: Brigham and Women's Hospital (Other); NYU Langone Health (Other); University of Pennsylvania (Other); Harvard Medical School (HMS and HSDM) (Other); New York University (Other)
Responsible Party: Sponsor
Other Study IDs: 202110921
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Psoriatic Arthritis; Psoriasis; Psoriatic Conditions; Dermatologic Disease; Rheumatologic Disease; Psoriatic Nail; Plaque Psoriasis; Joint Pain; Dactylitis
Keywords: Psoriasis; Psoriatic Arthritis; Psoriatic Disease; Health app research; mHealth research; Mobile health research
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Skin Diseases; Collagen Diseases; Arthralgia | interventions — Walking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Participants with Psoriasis: People who report a diagnosis of Psoriasis. Participants are invited via the Psorcast mobile application to complete the following assessments: Participant self-assessment surveys, skin assessments (Psoriasis Area Draw and Psoriasis Area Photo) and musculoskeletal assessments (Finger/Toe Photos, Joint Count, Digital Jar Open, 30s Walk).
  Interventions: Behavioral: Participant self-assessment surveys; Behavioral: Psoriasis Draw; Behavioral: Psoriasis Area Photo; Behavioral: Finger and Toe Photos; Behavioral: Digital Jar Open; Behavioral: 30 Second Walk; Other: Psorcast mobile application
- Participants with Psoriatic Arthritis: People who report a diagnosis of Psoriatic Arthritis. Participants are invited via the Psorcast mobile application to complete the following assessments: Participant self-assessment surveys, skin assessments (Psoriasis Area Draw and Psoriasis Area Photo) and musculoskeletal assessments (Finger/Toe Photos, Joint Count, Digital Jar Open, 30s Walk).
  Interventions: Behavioral: Participant self-assessment surveys; Behavioral: Psoriasis Draw; Behavioral: Psoriasis Area Photo; Behavioral: Finger and Toe Photos; Behavioral: Digital Jar Open; Behavioral: 30 Second Walk; Other: Psorcast mobile application
- Participants without Psoriasis or Psoriatic Arthritis: People who report no prior diagnosis of Psoriasis or Psoriatic Arthritis. Participants are invited via the Psorcast mobile application to complete the following assessments: Participant self-assessment surveys, skin assessments (Psoriasis Area Draw and Psoriasis Area Photo) and musculoskeletal assessments (Finger/Toe Photos, Joint Count, Digital Jar Open, 30s Walk).
  Interventions: Behavioral: Participant self-assessment surveys; Behavioral: Psoriasis Draw; Behavioral: Psoriasis Area Photo; Behavioral: Finger and Toe Photos; Behavioral: Digital Jar Open; Behavioral: 30 Second Walk; Other: Psorcast mobile application

INTERVENTIONS:
Behavioral: Participant self-assessment surveys — At enrollment, participants are asked to complete a baseline health history, family history, and a participant-reported symptom inventory.
Behavioral: Psoriasis Draw — Participants are asked to draw the location and size of psoriasis they currently experience. Participants are provided a body template onto which they can draw on their screen. Investigators estimate the percentage of body area affected.
Behavioral: Psoriasis Area Photo — Participants are asked to take a picture of a representative psoriasis plaque and indicate the location of the plaque. They are asked to take a picture of the same area over time. The investigators are developing computer vision algorithms to assess the plaque.
Behavioral: Finger and Toe Photos — Participants are asked to take pictures of the back of each hand and the top of each foot. These photos can be used to assess finger and toe swelling as well as psoriatic nail involvement. The investigators are developing computer vision algorithms to assess psoriatic nail involvement and digit swelling.
Behavioral: Digital Jar Open — Participants are asked to internally and externally rotate the phone as it rests on a flat surface. Participants perform each direction (internal and external) and each arm (left and right) in turn. Gyroscope sensors measure the degree of rotation.
Behavioral: 30 Second Walk — Participants are asked to walk in a straight line for 30 seconds. Gait is measured by gyroscope and accelerometer sensors. The investigators examine step-dependent and sequence-dependent features from these sensors. The investigators apply feature selection and classifier algorithms to analyze these data.
Other: Psorcast mobile application — Participants complete all described behavioral interventions via a dedicated iPhone app, Psorcast.

SUMMARY:
The purpose of this study is to understand variation in the symptoms of psoriasis and psoriatic arthritis using simple, scalable smartphone-based measurements. This study uses an iPhone app to record these symptoms through questionnaires and sensors.

DETAILED DESCRIPTION:
Psoriatic disease exhibits a spectrum of symptoms and can transition from psoriasis (PsO), largely affecting the skin, to psoriatic arthritis (PsA) involving widespread musculoskeletal inflammation. Early detection of the PsO-to-PsA transition and rapid administration of effective treatment is essential, as a delay in diagnosing PsA by as little as 6 months can lead to irreversible joint damage. This "ticking clock" paradigm drives the need for frequent monitoring and effective therapeutic intervention as early as possible to attenuate or possibly prevent disease progression. Using a suite of smartphone-based measurements in an app called Psorcast (psoriasis forecasts), we aim to aggregate weekly, symptom measurements from participants in a remote, longitudinal observational study to map the trajectories of treatment response and disease progression. In this study, we will explore measurements of psoriatic disease activity at least an order of magnitude more frequently (weekly vs. quarterly) than standard clinical practice or clinical trial designs. This study is not meant to provide a medical diagnosis, treatment, or medical advice. It is meant to provide a scalable, inexpensive, non-invasive and frequent measure and tracking of psoriasis and psoriatic arthritis for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 and older who consent to participate in the study
* Own a compatible iPhone or iPod Touch device running iOS 12.2 or above
* Be able to read and understand an official language of the country of participation

Exclusion Criteria:

* Age 17 years or younger
* Not a resident of the a country where the app is approved for use
* Not have a personal (i.e., not shared) iPhone (4s or newer running iOS 8.0 or later)
* Not be able to read and understand an official language of the country of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with a compatible iPhone or iPod Touch who consent to particpate
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Results of participant self-assessment surveys | Through study completion, an average of 2 years
  Results of participant self-assessment surveys will be analyzed using descriptive statistics. These results may also be compared with other intervention results.
Body surface area and location from the Psoriasis Draw assessment | Through study completion, an average of 2 years
  The investigators will quantify body surface area and psoriasis area hotspots across the cohort. These results may also be compared with other intervention results.
Computer vision features from Psoriasis Area Photo assessment | Through study completion, an average of 2 years
  The investigators apply visual processing and classifier algorithms to analyze the images from the Psoriasis Area Photo assessments. These results may also be compared with other intervention results.
Computer vision features from Finger/Toe Photos | Through study completion, an average of 2 years
  The investigators apply visual processing and classifier algorithms to segment nails and joints from hand and foot photos. These results may also be compared with other intervention results.
Gyroscope and accelerometer sensor measurements from Digital Jar Open assessment | Through study completion, an average of 2 years
  The investigators examine rotational features from gyroscope and accelerometer sensors. The investigators apply feature selection and classifier algorithms to analyze these data. These results may also be compared with other intervention results.
Gyroscope and accelerometer sensor measurements from 30-sec Walk assessment | Through study completion, an average of 2 years
  The investigators examine step-dependent and sequence-dependent features from gyroscope and accelerometer sensors. The investigators apply feature selection and classifier algorithms to analyze these data. These results may also be compared with other intervention results.
Quantification and distribution of self-reported painful joints | Through study completion, an average of 2 years
  The investigators will quantify the self-reported painful joints and, in particular, compare to measurements from the 30-sec Walk and Digital Jar Open to identify correlations. These results may also be compared with other intervention results.

SECONDARY OUTCOMES:
App usage data for assessment of participant engagement | Through study completion, an average of 2 years
  App usage data is used to gauge participant engagement throughout the study period. These results may also be compared with other intervention results.

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Sieberts, Ph.D, Principal Investigator — Sage Bionetworks; Jose Scher, MD, Principal Investigator — NYU Langone Medical Center; Joseph Merola, MD, MMSc, Principal Investigator — Brigham and Women's Hospital & Harvard Medical School
Locations (1):
- Sage Bionetworks, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the de-identified data from participants who opt-in to data sharing during enrollment and consent.
Supporting Information: Analytic Code

REFERENCES:
- [Background] DE Webster, RH Haberman, LM Perez Chada, M Tummalacherla, A Tediarjo, V Yadav, E Chaibub Neto, W MacDuffie, M DePhillips, E Sieg, S Catron, C Grant, W Francis, M Nguyen, M Yussuff, RL Castillo, D Yan, AL Neimann, SM Reddy, A Ogdie, A Kolivras, MR Kellen, LM Mangravite, SK Sieberts, L Omberg, JF Merola, JU Scher medRxiv 2022.04.13.22273676; doi: https://doi.org/10.1101/2022.04.13.22273676
- See also: Psorcast Study Website — http://www.psorcast.org
- See also: Study App (App Store) — https://apps.apple.com/us/app/psorcast/id1473504102